CLINICAL TRIAL: NCT00804596
Title: Labeling Comprehension and Performance Evaluation of the Apollo Blood Glucose Monitoring System With Capillary Blood [Commercial Name is CONTOUR® USB]
Brief Title: Evaluation of Labeling Comprehension and Performance of a New Blood Glucose Meter System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2008-18
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2010-03-09 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with diabetes (Other): Subjects with diabetes use a new blood glucose monitoring system with subject capillary blood.
  Interventions: Device: Apollo Blood Glucose Monitoring System

INTERVENTIONS:
Device: Apollo Blood Glucose Monitoring System — Subjects with diabetes were rated for success in performing tasks with a new blood glucose monitoring system (BGMS). Also, subjects and healthcare professionals (HCPs) used the new blood glucose monitoring system with subject capillary blood. All blood glucose results were compared to a laboratory glucose method - Yellow Springs Instrument(YSI) Analyzer.
  Other Names: Commercial name is CONTOUR® USB

SUMMARY:
The purpose of the study was to evaluate the acceptability of product user guides for untrained subjects and to evaluate the performance of the system with lay users and healthcare providers (HCPs).

DETAILED DESCRIPTION:
The study evaluated the acceptability of product labeling for performing blood glucose testing with the new blood glucose meter system (BGMS) and for using meter features. Sections of the User Guide and Quick Reference Guide that gave instruction on performing a blood glucose test and operating system features were evaluated, including instructions on connectivity of the system with a computer, meter setup, glucose trends display, and other system features. The study also evaluated the performance of the blood glucose meter system (BGMS) in the hands of subjects and healthcare professionals using capillary blood. Subjects and healthcare professionals provided feedback about the BGMS and its features. Some subjects took the system home to evaluate the robustness of the BGMS.

ELIGIBILITY:
Inclusion Criteria:

* Have type 1 or type 2 diabetes
* Be at least 18 years of age but have not reached their 76th birthday, with approximately 50% (+10%) being less than 55 years of age, at time of consent
* Be willing to complete all study procedures
* Be routinely testing their blood sugar at home (at least once per day)
* Be able to speak, read, and understand English and understand the Informed Consent document
* Be able to read the labeling instructions
* Own or operate a computer for personal or professional use beyond that for email correspondence. Subjects will not have to use their personal computer for the study, but computer use will be required.

Exclusion Criteria:

* Minors <18 years of age and adults >75 years of age
* Pregnancy
* Physical (dexterity), visual, or neurological impairments that would make the person unable to perform testing with the BGMS
* Disorders in the fingertip lancing areas
* Acute or chronic infections, particularly skin infections
* Infection with a blood borne pathogen
* Taking prescription anti-coagulants or having clotting problems that may prolong bleeding. Taking aspirin daily (81mg or 325 mg) is not reason for exclusion
* Hemophilia or any other bleeding disorder
* Having a condition which, in the opinion of the Principal Investigator or designee, would put the person at risk or seriously compromise the integrity of the study
* Working for a competitive medical device company

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cuddihy, MD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 subjects signed informed consents but did not meet inclusion/exclusion criteria so were not considered enrolled in the study.
Groups:
- Subjects With Diabetes: Subjects with diabetes and healthcare professionals (HCPs) use a new blood glucose monitoring system with subject capillary blood.
Period: Overall Study
Arm/Group | Subjects With Diabetes
Started | 74
Completed | 74
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 74

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Rated as <=3 (Comprehension of Labeling)
Description: Study staff rated participants on their success at performing Blood Glucose (BG) testing and other system features after subjects read product labeling. The rating scale was:
  1. Successful in performing tasks correctly without assistance
  2. Successful after being referred to user instructions
  3. Successful after verbal assistance or review of part of user instructions (Similar to review of a specific function during a Customer Service call.)
  4. Unsuccessful (Incorrectly performed part of the testing regimen or required intervention by study staff.)
Time Frame: 1-2 hours
Population: per protocol
Measure: Number; unit: percentage of participants
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 74
percentage of participants
  Perfom blood glucose measurement | 100
  Connect meter to computer via USB port | 100
  Select 'Before'/"After' meal in Autolog feature | 100
  Access electronic user guide on Apollo meter | 100
  Set date/time to current by selecting Y at prompt | 100
  Remove meter from computer | 100
  Perform simulated BG test using control solution | 100
  Turn on test strip port light (n=73) | 100
  Access and review Logbook, Reports, and Summary | 100
  Access and review Blood Sugar Trends | 100
  Understand data for Before/After Meal and 14day | 100
  Understand Average glucose value | 100
  Understand BG number within target range | 100
  Understand BG number above target range | 100
  Understand BG number below target range | 100
  Was able to turn meter off (n=73) | 100
  Understand Apollo has no replaceable batteries | 100
  Able to charge via USB port and verify charging | 100
  Able to set date and time formats (n=73) | 100
  Able to change 'Before Meal' target range(n=73) | 100

2. Secondary Outcome: Number of Capillary Blood Results Within +/- 15mg/dL or +/- 20% of Laboratory Glucose Method
Description: Subjects with diabetes and healthcare professionals (HCPs) used a new Blood Glucose Monitoring System (BGMS) with subject capillary blood. The BGMS has programmed algorithms to provide results equivalent to either serum/plasma or whole blood glucose methods; this study evaluated results equivalent to plasma lab methods. All results were compared to a lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG results were obtained in duplicate from subjects using three lots of Contour Blood Glucose strips, evenly distributed among the subjects.
Time Frame: 1-2 hours
Population: Since each subject provided two blood glucose (BG) meter results, 2x74 (or 148) subject BG test results were possible. For each subject blood sample, a healthcare professional (HCP) provided two BG meter results so that 2x74 (or 148) BG results were possible for HCP test results.
Measure: Number; unit: Number of Duplicate Results (n=74x2)
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 74
Number of Duplicate Results (n=74x2)
  Subjects: Test Results (n=148) | 146
  HCPs: Test Results (n=148) | 143

ADVERSE EVENTS:
Arm/Group | Subjects With Diabetes
Serious Adverse Events (participants affected / at risk) | 0/74
Other Adverse Events (participants affected / at risk) | 4/74
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Diabetes (N=74)
Cold or flu-like symptoms during the home-use portion of the study (General disorders) | 4 (4) — Subjects reported cold or flu-like symptoms during the home-use portion of the study. (Unrelated)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less